CLINICAL TRIAL: NCT01705327
Title: Fox Investigation for New Discovery of Biomarkers (BioFIND)
Brief Title: Fox Investigation for New Discovery of Biomarkers
Acronym: BioFIND
Status: Completed | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: BioFIND
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2013-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; Biomarkers; Neurodegenerative disorder
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid (CSF), whole blood, DNA, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease Subjects
- Healthy Control Subjects

SUMMARY:
This is an observational, multi-center study to assess clinical features and biologic biomarkers in Parkinson's disease (PD) patients compared to healthy controls (HC). The primary objective of this study is to discover clinical and biologic markers of PD for use in clinical trials of disease-modifying therapies.

DETAILED DESCRIPTION:
BioFIND is a two-year observational clinical study designed to discover and verify biomarkers of Parkinson's disease (PD). BioFIND is collecting clinical data and biospecimens, including blood and cerebrospinal fluid (CSF), in a population of 120 well-defined, moderately advanced PD subjects and 120 healthy controls.

BioFIND will follow standardized data acquisition protocols to ensure that tests and assessments conducted at multiple sites can be pooled. Data and samples acquired from study participants will enable the development of a comprehensive Parkinson's database and biorepository, which will be available to the scientific community to conduct research on novel PD biomarkers.

ELIGIBILITY:
Inclusion Criteria (PD Subjects):

* Subjects must have bradykinesia and rigidity.
* Current or history of well documented resting tremor.
* Unilateral onset or persistent asymmetry.
* A well established response to dopaminergic agents including the presence of levodopa induced dyskinesia for at least 3 years according to treating physician's judgment.
* Subject has progressive PD of 5 to 18 years of duration from the onset of symptoms.
* Male or female age of onset of PD 50 to 70 by history. Current ages would range from 55 to 93 based on #5 and #6 requirements.
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* Willing and able to comply with scheduled visits, required study procedures and laboratory tests.

Exclusion Criteria (PD Subjects):

* Family history of PD in first degree relatives.
* Ashkenazi Jewish subject (defined as all 4 grandparents being Ashkenazi Jewish) will be excluded because of the high likelihood of genetic forms of PD (LRRK2) and GBA), unless these have been already excluded by genetic testing.
* Has others serious neurological disorders (clinically significant stroke, brain tumor, hydrocephalus, epilepsy, other neurodegenerative disorders, encephalitis, repeated head trauma).
* Has early severe autonomic involvement. Symptomatic orthostatic, hypotension or urinary incontinence within one year of onset of disease symptom.
* Current treatment with anticoagulants (e.g., Coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
* Use of investigational drugs or devices within 60 days prior to baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).
* Has lower body predominant symptoms.
* Has supra-nuclear gaze palsy, CG sign, corticospinal track signs.

Inclusion Criteria (HC Subjects):

* Male or female age 55 to 93 years at visit 1.
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* Willing and able to comply with scheduled visits, required study procedures and laboratory tests.

Exclusion Criteria (HC Subjects):

* Family history of PD in first degree relatives.
* Ashkenazi Jewish subject (defined as all 4 grandparents being Ashkenazi Jewish) will be excluded because of the high likelihood of genetic forms of PD (LRRK2) and GBA), unless these have been already excluded by genetic testing.
* Has other serious neurological disorders (clinically significant stroke, brain tumor, hydrocephalus, epilepsy, other neurodegenerative disorders, encephalitis, repeated head trauma).
* Has a history of cancer, autoimmune disorder, liver disease, or hematological disorders within the past 5 years.
* Has early severe autonomic involvement: symptomatic orthostatic hypotension or urinary incontinence within one year of onset of disease symptom.
* Current treatment with anticoagulants (e.g., Coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
* Use of investigational drugs or devices within 60 days prior to baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).
* MoCA score <26.

Ages: 55 Years to 93 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease and healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
No primary outcome measure | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldman, MD, MS, Principal Investigator — Rush University Medical Center; Roy Alcalay, MD, MS, Principal Investigator — Columbia University; Claire Henchcliffe, MD, D. Phil, Principal Investigator — Well Cornell Medical Center; Tao Xie, MD, PhD, Principal Investigator — University of Chicago; Paul Tuite, MD, Principal Investigator — University of Minnesota Medical Center; Un Jung Kang, MD, Study Chair — University of Chicago; Cindy Casaceli, MBA, Principal Investigator — Clinical Trial Coordinating Center, University of Rochester; Penelope Hogarth, MD, Principal Investigator — Oregon Health and Science University; Samuel A. Frank, MD, Principal Investigator — Boston Medical Center; Amy Amara, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Cornell University Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Derived] Paslawski W, Svenningsson P. Elevated ApoE, ApoJ and lipoprotein-bound alpha-synuclein levels in cerebrospinal fluid from Parkinson's disease patients - Validation in the BioFIND cohort. Parkinsonism Relat Disord. 2023 Nov;116:105765. doi: 10.1016/j.parkreldis.2023.105765. Epub 2023 Jul 12. PMID 37479568